CLINICAL TRIAL: NCT05915715
Title: Comparative Effects of McGill Stabilization Exercises and Proprioceptive Neuromuscular Facilitation Technique on Pain, Range of Motion and Functional Disability in Chronic Non-specific Low Back Pain
Brief Title: McGill Stabilization Exercises VS Proprioceptive Neuromuscular Facilitation Technique in Chronic Non-specific LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0124
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Chronic Non-specific Low Back Pain
Keywords: Non-specific Low back pain, McGill, Paraspinal muscles

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McGill stabilization exercise (Experimental): The patients performed the corresponding exercises 3 days a week and 10 repetitions of each exercise for a period of 6 weeks and a rest interval of 2 minutes between exercises
  Interventions: Other: McGill stabilization exercise
- Proprioceptive neuromuscular facilitation technique (Experimental): The total duration of RS will be of approximately 33 minutes
  Interventions: Other: Proprioceptive neuromuscular facilitation technique

INTERVENTIONS:
Other: McGill stabilization exercise — McGill Curl Up Lie down on your back.
  The Side Bridge Lie on your side.
  The Bird Dog.
  Arms: McGill stabilization exercise
Other: Proprioceptive neuromuscular facilitation technique — . The patient is in sitting position and faces the physical therapist. The RST program consisted of alternating (trunk flexion-extension) isometric contractions against resistance for 10 seconds, with no motion intended. Subjects performed 3 sets of 15 repetitions at maximal resistance provided by the same physical therapist. Rest intervals of 30 seconds and 60 seconds were provided after the completion of 15 repetitions for each pattern and between sets, respectively.
  Arms: Proprioceptive neuromuscular facilitation technique

SUMMARY:
Non-specific chronic low back pain (NS-CLBP) is defined as lumber pain persisting for longer than three months, in absence of a suspected pathology or any specific cause. A specific diagnosis of low back pain cannot be obtained in approximately 80% patients with low back pain, indicating that patients with low back pain are often diagnosed with non-specific low back pain and these are the majority of the individuals with low back pain that present to physiotherapy In other cases the cause may be a minor problem with a disc between two spinal bones (vertebrae), or a minor problem with a small facet joint between two vertebrae. There may be other minor problems in the structures and tissues of the lower back that result in pain. Objective of this study is to compare the effects McGill stabilization exercises and proprioceptive neuromuscular facilitation technique on pain, range of motion and functional disability in chronic non-specific Low back pain.

DETAILED DESCRIPTION:
Low back pain (LBP) is one of the commonest musculoskeletal disorders and one of the most demanding ones in cost of care and medical attention. It was stated earlier that 70% of adults would experience LBP at least once over their lifespan. Furthermore, over 80% of such patients report recurrent episodes. The worldwide point prevalence of low back pain (acute, subacute and chronic) was 7.83% in 2017, with 577 million people affected at any one time. In 2017, low back pain was responsible for around 65 million years lived with disability, representing a deterioration of about 17.5% since 2007 mainly owing to population growth and ageing, with the greatest increase recorded for low-income and middle-income countries. People more often leave their job because of low back pain than diabetes, hypertension, neoplasm, asthma, heart and respiratory disease combined. A sedentary lifestyle with a lack of physical activity results in the loss of muscle power and strength and can be a predictor of LBP leading to recurrent LBP. Non-specific chronic low back pain (NS-CLBP) is defined as lumbar pain persisting for longer than three months, in absence of a suspected pathology (red flag conditions such as e.g. tumor, infection or fracture).Patients commonly have limited range of motion and dis-coordination in the function of various body parts due to pain. Nonspecific LBP is described as pain that has no specific pathology as infection, neoplasm, etc.; rather, it might develop for mechanical reasons. It is characterized by heavy pain worsening with exertion, especially in the afternoon, and reliving with rest. Moreover, the application of faulty ergonomic principles may be a cause of LBP or worsen its symptoms. Chronic LBP is associated with histomorphologic and structural changes in the paraspinalis muscles. These back muscles are smaller, contain fat, and show a degree of atrophic changes in select muscle fibers. Therefore, the lumbar paraspinalis muscles are weak with excessive fatigability. Furthermore, poor coordination of the paraspinalis muscles has been associated with chronic LBP. These contribute to a vicious cycle of LBP and deconditioning syndrome. One type of NSCLBP is continuing and recurrent primarily nociceptive CLBP due to vertebral joint overload subsequent to functional instability of the lumbar spine. This condition may occur due to disruption of the motor control system to the key stabilizing muscles in the lumbar spine, particularly the lumbar multifidus muscle (MF).Traditionally, treatment of CLBP has focused on analgesia and activity restriction. However, this treatment is ineffective and can even be harmful, generating distrust among patients and frustration towards PHCPs. Most guidelines agree on the first line of care in case of acute episode: advice, reassurance and encouragement to engage in light physical activity. When second-line treatment is needed, a range of therapeutic interventions (pharmacological and physiotherapy) for acute NSLBP are available. Patients with CLBP usually have more comorbidity and impose greater economic burdens to the society than those without CLBP. Recent research shows that the number of people with disabilities caused by chronic LBP has increased by 54% in the last 30 years.Thus, LBP poses substantial challenges for the medical system, creates socioeconomic issues for working-age adults, and levies a severe medical burden on individuals and society.

Nonspecific CLBP pain is associated with major depression, decreased productivity, disability, and reduced life quality. Therefore, there is an urgent need for research to better understand the underlying mechanisms that cause and sustain nonspecific CLBP and guide effective treatments. Exercise is an effective, non-pharmacologic treatment for chronic LBP, and most clinical practice guidelines recommend exercise as first-line treatment for chronic LBP. However, there is limited evidence about which exercise is best and the long-term effects of different exercise-based treatments.Proprioceptive neuromuscular facilitation (PNF) training has been recommended for sensorimotor control training as well as for stimulating lumbar muscle proprioception. Basic procedures, such as rotational patterns of movement and different techniques, including rhythmic stabilization, dynamic reversals, combination of isotonics, repeated contractions, and contract-relax, can be applied to improve flexibility, muscle strength, and movement. Thus, the concept of PNF is to enhance joint coordination, muscle strength, movement control, stability, and mobility. Its main objective is to reach the highest possible functional level. To achieve the highest functional level, therapists apply motor control and motor learning principles when using PNF. Exercises improve muscle strength, flexibility, endurance, and ability to perform life activities. Proprioceptive neuromuscular facilitation (PNF) involves stretching, resisted movements which improves muscle disharmony, atrophy, and joint movement limitation. Lumbar stabilization exercises (LSE) develop the awareness of muscle contraction and control from simple to complex patterns. Both exercises are effective individually in chronic low back pain patients. This study was conducted to find out which technique is better.

ELIGIBILITY:
Inclusion Criteria:

1. 20-40years
2. Both Genders.
3. Mild to moderate back pain with NPRS pain score of between 2/10- 6/10.
4. Chronic low back pain for more than 3 months.
5. No radiating pain below the gluteal fold.

EXCLUSION CRITERIA

1. Diagnosed with disc herniation
2. lumber canal stenosis
3. spondylolysis,
4. Lumbar radiculopathy
5. Lumbar vertebral fracture
6. Any referred pain below gluteal fold or neurological involvement in lower limbs
7. Participants who had undergone surgery for lumbopelvic surgery, abdominal, shoulder and lower limb surgery.
8. Pregnancy.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
1. Numerical Rating Scale (NPRS) | [Time Frame: 6th week]
  Numeric Rating Scale (NPRS) is most frequently used instruments to measure pain intensity in neck pain .The 11-point numeric with 0 representing No pain, 1-3 representing Mild Pain (nagging, annoying, interfering little with ADLs), 4-6 representing Moderate Pains (interferes significantly with ADLs), 7-10 representing Sever Pain (disabling, unable to perform ADLs)
2. Bubble Inclinometer | [Time Frame: 6th week]
  The spinous process of the 1st sacral vertebra and the 12th thoracic vertebra were considered as reference points for measuring the range of motion in bending forward and backward. The spinous process of the 12th thoracic vertebra was considered as reference point for measuring the range of motion of lumbar side flexion. Two bubble inclinometers were used simultaneously for measuring the lumbar range of motion when bending forward (in the standing position), and one bubble inclinometer for measuring the lumbar range of motion for back extension (in the standing) and side flexion (in the standing position).The actual ranges of motion of lumbar area when bending forward and backward were calculated by subtracting the number (degree) obtained by the lower inclinometer from the number (degree) obtained by the upper inclinometer
3. Modified Oswestery Disability Index (MODI) | [Time Frame: 6th week]
  For patients with low back pain, the Oswestry Disability Index (ODI) is a well-recognized and widely used patient reported health questionnaire and outcome measure. It is a self-rating questionnaire comprised of a series of ten sections, each with six statements describing functional impairment in a variety of activities of daily living including: personal care, lifting, sitting, standing, walking, sleeping, sex life, social life and travelling, as well as the intensity of pain and its response to analgesia. The six statements are scored from 0-5 and responses are added to give a total score out of a maximum possible score of 50 (or 45 if the question on sex life is omitted).
  This score can subsequently be categorized in to five levels of increasing disability

SECONDARY OUTCOMES:
ROM lumber spine (flexion) | [Time Frame: 6th week]
  To measure total flexion ROM, the spinous process of T12 is identified and marked. The inclinometer is centered over the mark at T12 and zeroed. The patient is instructed to bend forwards as far as possible without bending the knees. The ROM value on the inclinometer is recorded for total flexion.
ROM lumber spine (side flexion) | [Time Frame: 6th week]
  To measure side bending ROM, the inclinometer is placed just above the mark at T12 parallel to the axis of the spinal column and zeroed. The patient is instructed to lean over to the right or left as far as possible with the fingertips reaching as far down the side of the thigh, and the ROM value on the inclinometer is recorded.
ROM lumber spine (extension) | [Time Frame: 6th week]
  To measure extension, the inclinometer is centered over the mark at T12, and the inclinometer is zeroed. The patient is instructed to bend backwards as far as possible without bending his knees, and the ROM value for extension was recorded.
ROM lumber spine (rotation) | [Time Frame: 6th week]
  Patient is standing and forward flexed spine positioned in neutral rotation place bubble inclinometer on s1 and T12 ask patient to rotate and measure the reading with both inclinometers first set to zero.

CONTACTS AND LOCATIONS:
Overall Officials: Sana Hafeez, PhD*, Principal Investigator — Riphah International University Lahore Campus
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fouda KZ, Dewir IM, Abdelsalam MS. Effects of proprioceptive neuromuscular facilitation techniques in treating chronic nonspecific low back pain patients. Physiotherapy Quarterly. 2021;29(2):32-7.
- [Background] Gianola S, Bargeri S, Del Castillo G, Corbetta D, Turolla A, Andreano A, Moja L, Castellini G. Effectiveness of treatments for acute and subacute mechanical non-specific low back pain: a systematic review with network meta-analysis. Br J Sports Med. 2022 Jan;56(1):41-50. doi: 10.1136/bjsports-2020-103596. Epub 2021 Apr 13. PMID 33849907
- [Background] Dal Farra F, Risio RG, Vismara L, Bergna A. Effectiveness of osteopathic interventions in chronic non-specific low back pain: A systematic review and meta-analysis. Complement Ther Med. 2021 Jan;56:102616. doi: 10.1016/j.ctim.2020.102616. Epub 2020 Nov 13. PMID 33197571
- [Background] Suh JH, Kim H, Jung GP, Ko JY, Ryu JS. The effect of lumbar stabilization and walking exercises on chronic low back pain: A randomized controlled trial. Medicine (Baltimore). 2019 Jun;98(26):e16173. doi: 10.1097/MD.0000000000016173. PMID 31261549
- [Background] Russo M, Deckers K, Eldabe S, Kiesel K, Gilligan C, Vieceli J, Crosby P. Muscle Control and Non-specific Chronic Low Back Pain. Neuromodulation. 2018 Jan;21(1):1-9. doi: 10.1111/ner.12738. Epub 2017 Dec 12. PMID 29230905
- [Background] Garcia-Martinez E, Soler-Gonzalez J, Blanco-Blanco J, Rubi-Carnacea F, Masbernat-Almenara M, Valenzuela-Pascual F. Misbeliefs about non-specific low back pain and attitudes towards treatment by primary care providers in Spain: a qualitative study. BMC Prim Care. 2022 Jan 14;23(1):9. doi: 10.1186/s12875-021-01617-3. PMID 35172719
- [Background] Chang JR, Wang X, Lin G, Samartzis D, Pinto SM, Wong AYL. Are Changes in Sleep Quality/Quantity or Baseline Sleep Parameters Related to Changes in Clinical Outcomes in Patients With Nonspecific Chronic Low Back Pain?: A Systematic Review. Clin J Pain. 2021 Dec 22;38(4):292-307. doi: 10.1097/AJP.0000000000001008. PMID 34939973